CLINICAL TRIAL: NCT03172767
Title: The Relationship Between School Readiness and Sensory Processing Disorder in Preterm Preschooler
Acronym: Preterm
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Principal Investigator, Gazi University
Other Study IDs: 5461
Record Dates: First submitted 2017-05-26; First posted 2017-06-01 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2017-05

CONDITIONS: Sensory Deficit; Preterm Birth
Keywords: Preterm; Sensory processing; School Readiness
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm Preschoolers: Preterm children who haven't attend school.
- Term Preschoolers: Term children who haven't attend school.

SUMMARY:
The study aims investigate sensory processing disorders and school readiness in pre-school preterm children and the relationship between sensory impairment and school readiness

DETAILED DESCRIPTION:
A convenience of preterm and term preschoolers recruiting from Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation. Each group contains 30 children. First, sociodemographic information and histories of children are obtaining. Ages and contact information of the parents are recording. Prenatal and natal risk factors of the mothers are querying. Gestational ages and height, weight, and head circumferences of babies at birth are recording. Number of pregnancies, live births and abortions, type of delivery, multiple pregnancies for mothers as well as consanguinity between parents are asking. Marmara Primary School Readiness Scale is using to evaluate mental-language development, socio-emotional development, physical development, self-care skills,math skills, science skills, voice exercises, line exercises and labyrinths. Sensory profile caregiver questionnaire screen for the senses (sensory processing), adjustment (modulation), behavioral and emotional responses. . All examination wiil be finished in the same day.

ELIGIBILITY:
Inclusion Criteria:

* No neurological diagnosis
* gestational age < 37 weeks
* 60-78 months of age

Exclusion Criteria:

* Have a neurological diagnosis (such as cerebral palsy)
* Grade III or grade IV intraventricular hemorrhage
* Have undergone major surgery in neonatal period
* Mental retardation

Ages: 60 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm Preschoolers and Term Preschoolers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Marmara Primary School Readiness Scale | 45 minutes
  The application form includes math skills, science skills, voice exercises, line exercises and labyrinths; Development form; Mental-language development, socio-emotional development, physical development, self-care skills.

SECONDARY OUTCOMES:
Sensory profile caregiver questionnaire | 45 minutes
  The profile reveals the child's sensory appearance in terms of sensory search, emotional response formation, low endurance, oral tenderness, distractibility, weak perception, sensory sensitivity, activity level and fine motor / perceptual differences. In addition, the child evaluates the senses (sensory processing), adjustment (modulation), behavioral and emotional responses.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Study Chair — study chair
Locations (1):
- Gazı University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes